CLINICAL TRIAL: NCT06638281
Title: Reliability of the Incremental Shuttle Walk Test in University Students
Status: Completed | Type: Observational
Sponsor: Siirt University (Other)
Responsible Party: Principal Investigator, Yasemin ACAR, Research Assistant, Siirt University
Other Study IDs: 2024/05/01/06
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Incremental Shuttle Walk Test
Keywords: exercise tolerance; exercise test; Test-Retest Reliability; Reliability of Results

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the inter-rater and intra-rater reliability of the incremental shuttle walk test in university students.

DETAILED DESCRIPTION:
The incremental shuttle walk test (ISWT) is a valid and reliable field test developed to evaluate functional exercise capacity. This test requires the participant to walk up and down a 10 m course marked by two cones placed 9 m apart. The walking speed, determined by an audio signal, is slow at first, but gradually increases every minute.

Although validity and reliability studies have been conducted in different disease groups and healthy populations, there is no study evaluating the inter-rater reliability of the incremental shuttle walk test in healthy individuals. Our research aims to evaluate the inter-rater and intra-rater reliability of the incremental shuttle walk test in university students.For this purpose, undergraduate nursing students will be included in our research.ISWT will be administered to students by two different researchers on the same day. For test-retest reliability the ISWT will be administered again by the same researchers on a different day (retest).

ELIGIBILITY:
Inclusion Criteria:

* Being a student of Siirt University Faculty of Health Sciences, Nursing Department
* Being between the ages of 18-26
* Understanding and speaking Turkish

Exclusion Criteria:

* Having a systemic, orthopedic or neurological disease
* Participant wishes to withdraw from the study

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Siirt University Faculty of Health Sciences, Nursing Department students
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Incremental Shuttle Walk Test Results | At baseline and within 2-7 days after first assessment
  The number of completed shuttles will be recorded, and the total incremental shuttle walk distance (ISWD) will be calculated. Heart rate (HR), arterial blood pressure, saturation, perceived dyspnea, and fatigue according to the modified Borg scale will be assessed before, at the end of the test, and after a 5-min recovery.

SECONDARY OUTCOMES:
Age | Baseline
  Age in years
Weight | Baseline
  Weight (kg)
Height | Baseline
  Height (m)
Smoking Status | Baseline
  Smoking status will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin ACAR, Study Director — Siirt University
Locations (1):
- Siirt University, Siirt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No